CLINICAL TRIAL: NCT03403153
Title: Adaptation, Refinement, and Open Trial of Parent Training for Veterans With PTSD
Brief Title: Parenting Strength At Home- Parents Pilot
Acronym: PSAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D2421-R
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Results first posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Parenting Behaviors and PTSD Symptoms
Keywords: Parent-Child Relationship; military family; veterans health; stress disorders
MeSH Terms: conditions — Stress Disorders, Traumatic

STUDY DESIGN:
Intervention Model Description: This study is examining the feasibility and acceptability of an intervention to improve parent-child functioning. It will also conduct a preliminary test for movement in target outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pilot and Open Trial (Other): All Participants will complete the 8-week parenting support intervention and will provide satisfaction and acceptability ratings of the intervention. In the pilot trial, participants will make these ratings after each session, in the open trial the ratings will be made pre and post intervention.
  Interventions: Behavioral: SAHP

INTERVENTIONS:
Behavioral: SAHP — Aim 1: To obtain and incorporate expert clinician and Veteran feedback on credibility, acceptability, and satisfaction with the intervention to ensure Veteran-friendly intervention manual, materials, and processes. Aim 1 will be accomplished through two rounds of expert panel review of treatment/MIA manual and two rounds of pilot testing of the treatment for Veteran Feedback in 16 female and 16 male Veterans.
  Aim 2: To evaluate feasibility of study recruitment, retention, assessment procedures and proposed methods of the intervention. Preliminary examination of whether the intervention results in improvements to parenting behaviors, parenting satisfaction and overall family functioning.

SUMMARY:
The overall goal of this work is to adapt, refine, and conduct an open trial of a parent-training intervention for Veterans with posttraumatic stress disorder (PTSD) symptoms using feedback from Veterans, VA clinicians, and expert consultants as key stakeholders. PTSD symptoms are associated with parent-child functioning difficulties, which are also an important determinant of quality of life and functional recovery. This project will examine the feasibility and acceptability of an evidence-based group intervention to improve parenting behaviors, parenting satisfaction, and family functioning in Veteran parents with PTSD symptoms and who have children between the ages of 3 and 12.

This intervention is derived from an existing evidence-based intervention to improve Veteran relationship functioning (Strength at Home; SAH), and it is informed by the Cognitive Behavioral Theory of Interpersonal Functioning and the Military Family Attachment frameworks for the association between PTSD and family functioning problems. The intervention also includes a pre-treatment Motivational Interviewing Assessment (MIA) to assist Veterans in strengthening and building motivation to change their parenting behaviors. The goals and change talk identified in the pre-treatment MIA are then referred to throughout the treatment. Groups are gender-specific, meaning that the investigators will pilot the treatment in separate groups of women and men Veterans.

DETAILED DESCRIPTION:
Symptoms of posttraumatic stress disorder (PTSD) after deployment have been shown to adversely impact family and close relationship functioning, including parent-child relationships. About 31% of U.S. Veterans are parents to children under the age of 18. In addition, a study of over 100,000 records of Iraq and Afghanistan Veterans indicated those with dependent children were 40% more likely to carry a diagnosis of PTSD compared to those without children. Despite these large numbers and the known association between PTSD and parenting problems, there are no empirically validated parenting interventions within the VHA that address the unique needs of Veteran parents with PTSD, nor is there evidence that existing treatments for PTSD improve family functioning. This gap in both research and practice is significant given that parent-child functioning is a large component of recovery and reintegration into the community. Difficulties with parenting and the parent-child relationship are a vital influence on overall family functioning and quality of life. It follows logically that an intervention that improves parenting will have a significant downstream impact on overall family and close relationship functioning and the Veteran's quality of life.

This proposal will conduct the research necessary to adapt, refine, and conduct an open trial of Strength at Home - Parents (SAHP) - the new intervention incorporates the core clinical components of the empirically validated Strength at Home (SAH) interventions for improved family functioning among Veterans and targets key parenting behaviors and interpersonal relationship skills that can be impaired when a parent suffers from PTSD.

Given that parenting challenges are not typically addressed within VHA, one reason prior national pilot efforts may have had trouble with enrollment and retention is a failure to address motivation and goal setting at the outset. It can be difficult for clients to be ready to change a problem when few resources have historically been available to address it. Therefore this proposal will pilot the feasibility of including a pre-treatment Motivational Interviewing Assessment (MIA15) to assist Veterans with PTSD in strengthening and building motivation to change their parenting behaviors. The MIA can result in higher rates of treatment retention during the first 4 weeks of treatment compared to treatment as usual. Assessment approaches such as MIA that are personalized and collaborative have been shown to have a positive and clinically meaningful impact on treatment.

ELIGIBILITY:
Inclusion Criteria:

* English speaking and able to provide written informed consent
* Current parent to a child between the ages of 3 and 12.

  * If the parent has more than one child within the target group, they will choose one of their children to be the index child for the purposes of SAHP
  * Though we expect skills learned will translate to other children in the family
  * The child must reside with the Veteran or spend at least an average of two days per week with the Veteran
* Screen positive for elevated PTSD symptoms on the PTSD checklist for DSM 5 (PCL-5)

  * The PCL-5 is a 20 item self-report measure of PTSD symptoms in the past month. Items are rated on a 5 point Likert scale (0 = not at all, 4= extremely) and participants endorse symptoms based on "a very stressful experience."
  * Items are summed with higher scores reflecting greater symptomatology. The measure evidences good reliability (Internal consistency = .96; test-retest = .84), discriminant and convergent validity and takes 5-10 min. to complete
* Screen positive (above the 85th percentile) for parent-child functioning problems based on Parenting Stress Index- Short Form; PSI-SF

  * All three subscales and the total stress scale on the short-form are highly correlated with those on the long-form (.97-.99), and is expected to take respondents about 10 minutes to complete
  * The total stress scale can successfully differentiate between different levels of risk for parent-child functioning problems and has strong convergent validity. High Cronbach's alpha scores have been reported across all scales, ranging from .88 to .9584

Exclusion Criteria:

* Major neurocognitive disorder, including due to TBI

  * The adapted Ohio State Traumatic Brain Injury Identification Method (OSU TBI-ID), is a 3-5 min. clinician administered interview for lifetime history of TBI
  * The OSU TBI-ID is a recommended common data element by NIH and evidences good- excellent reliability and validity
  * The OSU TBI-ID will be used to identify severe TBI as defined as a score of 5
  * The participant's medical record may also be used for secondary verification in the case of TBI
  * For those scoring a 5, further referral and screening for comprehension ability will be recommended to determine exclusion (as the intent is to identify individuals who may not understand or comprehend study materials)
* Untreated/poorly managed psychosis or substance dependence

  * The Mini-International Diagnostic Interview (MINI), is a structured diagnostic interview that can be completed in less than 10 minutes
  * It is one of the most widely used diagnostic interviews and evidences psychometric properties that are like more complex and lengthier measures
  * The psychotic disorders and substance dependence subscales of the MINI will be used to screen for DSM-V criteria for current psychosis and substance dependence
  * Participants meeting the diagnostic criteria above will be asked about their current treatment and if needed, the PI (licensed clinical psychologist) will speak with them regarding their current treatment plan and interest in referrals
  * Those not engaged in treatment (diagnosis without ongoing medication management or psychotherapy) and/or evidencing need for referral to detox (e.g. symptoms of withdrawal), and/or evidencing symptoms that interfere with the intake assessment will be excluded and referred for treatment. Where possible, a warm handoff will always be provided
  * Participants will be welcomed back to the study once stabilized
* Current suicide risk

  * The Beck Depression Inventory-II (BDI-II), a 21-item self-report measure of depression symptoms (5 min. to complete), will be used to assess for suicide risk as defined as a score of 2 or more on the BDI-II suicide item
  * The BDI-II suicide item evidences a moderate correlation with the other scales of suicidal ideation in clinical samples, and has predictive validity
  * Follow-up risk-assessment will be provided by the PI who is a licensed clinical psychologist
  * Individuals will be eligible after crisis intervention has been received

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Groups are gender-specific, meaning that the investigators will pilot the treatment in separate groups of women and men Veterans.
Enrollment: 91 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzannah K. Creech, PhD, Principal Investigator — Central Texas Veterans Health Care System, Temple, TX
Locations (3):
- United States (3):
  - Austin Information Technology Center, Austin, TX, Austin, Texas
  - Central Texas Veterans Health Care System, Temple, TX, Temple, Texas
  - Central Texas Veterans Health Care System Waco VA Medical Center, Waco, TX, Waco, Texas

IPD SHARING:
Plan to Share IPD: No
Upon written request and IRB approval of sharing, final datasets will be made available in electronic computer readable form. Only de-identified non-PHI raw data will be shared.

REFERENCES:
- [Derived] Creech SK, Pearson R, Saenz JJ, Braciszewski JM, Riggs SA, Taft CT. Trauma-informed parenting intervention for veterans: A preliminary uncontrolled trial of Strength at Home-Parents. J Fam Psychol. 2023 Dec;37(8):1294-1302. doi: 10.1037/fam0001131. Epub 2023 Sep 14. PMID 37707465

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted between 3/01/2019 and 11/8/2019. Participants self-referred through study flyers or were recruited through letters sent to those veterans who met initial study eligibility based on medical record data.
Pre-assignment Details: Participants who were not retained at post-treatment cited logistical reasons for discontinuing in the study (e.g., work/school conflicts, travel time), and these participants mostly withdrew without attending any sessions.
Groups:
- SAHP Pilot: We aimed to recruit 20-32 participants across 2 male and 2 female (unyoked) pilot treatment groups. Although our recruitment target was partially constrained by pragmatic considerations, we believed that this sample size would allow us to test the feasibility of our recruitment methods and study procedures and give us sufficient quantitative and qualitative data on intervention reception. Ultimately, we recruited 12 female and 9 male Veterans.
- SAHP Open Trial: Strength at Home - Parents (SAHP) is a trauma-informed psychotherapy group that aims to improve parenting behaviors and overall parent-child and family functioning among U.S. military veterans with post-traumatic stress disorder (PTSD) symptoms. SAHP was developed to maximize ease of use by VA providers and accessibility for parents.
Period: Overall Study
Arm/Group | SAHP Pilot | SAHP Open Trial
Started | 21 (21 Veterans (42.0%) met initial eligibility criteria and completed an intake assessment.) | 53
Completed | 20 (20 participants (95.2%) elected to participate in treatment sessions.) | 47
Not Completed | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- SAHP Pilot; SAHP Open Trial: Strength at Home - Parents (SAHP) is a trauma-informed psychotherapy group that aims to improve parenting behaviors and overall parent-child and family functioning among U.S. military veterans with post-traumatic stress disorder (PTSD) symptoms. SAHP was developed to maximize ease of use by VA providers and accessibility for parents.
- Total: Total of all reporting groups
Arm/Group | SAHP Pilot | SAHP Open Trial | Total
Number analyzed (Participants) | 21 | 53 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 53 | 74
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 28 | 40
  Male | 9 | 25 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 10 | 10
  Not Hispanic or Latino | 0 | 43 | 43
  Unknown or Not Reported | 21 | 0 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 15 | 17
  White | 12 | 24 | 36
  More than one race | 7 | 10 | 17
  Unknown or Not Reported | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Client Satisfaction Questionnaire-8 (CSQ; Attkisson & Greenfield, 2004)
Description: The Client Satisfaction Questionnaire-8 (CSQ) assesses acceptability post-treatment. Eight items are scored on a 4-point scale inquiring about quality of services, treatment satisfaction, and willingness to recommend the treatment to others. Ratings are summed, with higher scores representing greater acceptability ratings (possible range 4-32). This measure is commonly used in both clinical trials and program evaluation, and has been shown to correlate with treatment attendance and outcomes. It takes approximately three minutes to complete. Evaluations of the measure found it to be reliable, with high coefficient alphas (.83-.93) to support internal consistency, and that it evidences positive construct validity with other measures of satisfaction. Where available, mean CSQ ratings can also be compared against norms from other studies in similar populations.
Time Frame: 8 weeks
Population: This measure given only in the Pilot trial.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- SAHP Pilot: All participants in the open trial and pilot received the intervention.
Arm/Group | SAHP Pilot
Number analyzed (Participants) | 21
score on a scale | 29.9 [4 to 32]

2. Primary Outcome: Strength at Home Parents Specific Satisfaction Questionnaire
Description: Measure was designed for this study and administered after each session to assess satisfaction with session components, overall session content, and homework. Sample questions include "The group exercise on child attachment was useful in understanding my child's behavior" and "The number of take home practice assignments is reasonable". Items are scored on a 9-point scale and averaged (range 0 - 8) with higher scores representing greater treatment satisfaction. Additional qualitative feedback was obtained using open-ended questions.
Time Frame: 8 weeks
Population: Only participants in the pilot completed this measure
Measure: Mean (Full Range); unit: score on a scale
Groups:
- SAHP Pilot: All participants in the pilot received the intervention.
Arm/Group | SAHP Pilot
Number analyzed (Participants) | 20
score on a scale | 6.65 [0 to 8]

3. Primary Outcome: The Credibility/Expectancy Questionnaire (CEQ; Devilly & Borkovec, 2000)
Description: Measure was administered after first and last session to assess participants perspectives on whether the intervention was logical and their expectations for the success of the intervention. There are 4 items scored on an 8-point scale (range 0-32), with higher scores representing greater credibility, and a reported mean score of 24.96 in standardization samples. Although CEQ session ratings were used to guide manual revisions, only CEQ scores at pre and post-treatment were evaluated for this report. The CEQ has high internal consistency and test-re-test reliability (Devilly & Borkovec, 2000).
Time Frame: 8 weeks
Population: Those in the pilot completed this measure.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | SAHP Pilot
Number analyzed (Participants) | 20
score on a scale
  1st session | 27.7 [0 to 32]
  last session | 28.9 [0 to 32]

4. Secondary Outcome: The Parenting Stress Index, 4th Edition (PSI; Abidin, 2012)
Description: Measure has 120 items scored on a 5-point scale, yielding a parent domain score, a child domain scale measuring stress related to parent and child characteristics respectively. These scale scores are combined (Summed) to yield a parenting stress index total score with higher scores reflecting greater stress. The PSI has high reliability coefficients, internal consistency, and test-retest reliability. The measure has been validated for use in various populations (Abidin, 2012). The range for the total score is 20-100.
Time Frame: 8 weeks
Population: Open trial subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SAHP Open Trial: All participants in the open trial and pilot received the intervention.
Arm/Group | SAHP Open Trial
Number analyzed (Participants) | 53
score on a scale
  Pre-treatment | 62 (8.95)
  post-treatment | 55.5 (7.95)
Statistical Analysis 1: Comparison: SAHP Open Trial; Test type: Other; p < 0.01, t-test, 1 sided

5. Secondary Outcome: The Family Assessment Device General Family Functioning Scale (FAD; Epstein, Baldwin, & Bishop, 1983)
Description: Measure is a 12-item measure on a 4 - point scale measuring general family functioning. Items are averaged (range 1 to 4), with higher scores reflecting impaired family functioning. The FAD has high Cronbach's alpha (.86), and split-half reliability (.83) (Byles, et al., 1988). Consistency between responses to the 12-item FAD, and related family variables provides validity evidence.
Time Frame: 8 weeks
Population: open trial outcomes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAHP Open Trial
Number analyzed (Participants) | 53
score on a scale
  pre-treatment | 2.17 (.5)
  post-treatment: number analyzed (Participants) | 47
  post-treatment | 1.86 (.6)
Statistical Analysis 1: Comparison: SAHP Open Trial; Test type: Other; p < .01, t-test, 1 sided

6. Secondary Outcome: The Pediatric Symptom Checklist (PSC; Jellinek, et al., 1986)
Description: Measure is a 35-item measure on a 3-point scale assessing parents' impressions of their child's psychosocial functioning. Scores range from 0 to 70, with higher scores reflecting greater psychosocial problems and impairment. The PSC converges with the Child Behavior Checklist, an established self-report measures of child psychosocial difficulties (Jellinek et al., 1986).
Time Frame: 8 weeks
Population: open trial subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAHP Open Trial
Number analyzed (Participants) | 53
score on a scale
  Pre-treatment | 20.6 (8.06)
  post-treatment: number analyzed (Participants) | 47
  post-treatment | 15.7 (8.12)
Statistical Analysis 1: Comparison: SAHP Open Trial; Test type: Other; p < .01, t-test, 1 sided

7. Secondary Outcome: The Parenting Scale Laxness Subscale
Description: Parental discipline practices were measured with the laxness and hostility subscales of the Parenting Scale (PS; Arnold et al., 1993). Scores are averaged with higher scores reflecting more dysfunctional parenting practices. Items are anchored by one effective and one ineffective discipline strategy rated on a 1 to 7 scale. The laxness scale is comprised of 11 items measuring permissive, inconsistent discipline e.g. "If my child gets upset when I say 'no': I back down and give in to my child (1)… I stick to what I said (7)." The overreactivity scale measures use of emotional, harsh discipline such as "When my child misbehaves I spank, slap, grab, or hit my child... never or rarely (1) …. most of the time (7)." Adequate internal consistency and reliability have been demonstrated, and the scale correlates well with observational measures of dysfunctional discipline and child misbehavior (Arnold et al. 1993).
Time Frame: 8 weeks
Population: open trial subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAHP Open Trial
Number analyzed (Participants) | 53
score on a scale
  pre-treatment | 2.68 (1.14)
  post-treatment: number analyzed (Participants) | 47
  post-treatment | 2.38 (.93)
Statistical Analysis 1: Comparison: SAHP Open Trial; Test type: Other; p < .01, t-test, 1 sided

8. Secondary Outcome: Beck Depression Inventory-II (BDI-II; Beck et al. 1996)
Description: Measure is a 21-item measure on a 4-point scale assessing depression symptom severity. Scores range from 0 to 63 with higher scores reflecting increased endorsement of depressive symptoms. The BDI-II has high internal consistency, good test-retest reliability (.94), and correlates highly with other interview-based measures of depression (Sprinkle et al., 2002).
Time Frame: 8 weeks
Population: open trial subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAHP Open Trial
Number analyzed (Participants) | 53
score on a scale
  Pre-treatment | 27.6 (13)
  Post-treatment: number analyzed (Participants) | 47
  Post-treatment | 21 (11.8)
Statistical Analysis 1: Comparison: SAHP Open Trial; Test type: Other; p < .01, t-test, 1 sided

9. Secondary Outcome: PTSD Checklist for DSM-5 (PCL-5; Weathers et al. 2013)
Description: Measure is a 20-item measure on a 5-point scale assessing PTSD symptom severity. Scores range from 0 to 80 with higher scores reflecting increased endorsement of PTSD symptoms. The measure has good internal consistency, test-retest reliability and convergent and discriminant validity (Blevins, et al., 2015). The PCL-5 is as sensitive to clinical change that occurs between pre-and post- treatment as golden standard interview-based measures of PTSD symptoms (Worthmann et al., 2016).
Time Frame: 8 weeks
Population: open trial subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAHP Open Trial
Number analyzed (Participants) | 53
score on a scale
  pre-treatment | 44.1 (16.1)
  post-treatment: number analyzed (Participants) | 47
  post-treatment | 35.5 (17.8)
Statistical Analysis 1: Comparison: SAHP Open Trial; Test type: Other; p < .01, t-test, 1 sided

10. Secondary Outcome: Parenting Stress Index Hostility Subscale
Description: as for outcome 7
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SAHP Open Trial
Number analyzed (Participants) | 53
units on a scale
  pre-treatment | 2.35 (1.25)
  post-treatment | 1.86 (.94)
Statistical Analysis 1: Comparison: SAHP Open Trial; Test type: Other; p < .01, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Two months.
Groups:
- Pilot Trial; Open Trial: All Participants will complete the 8-week parenting support intervention and will provide satisfaction and acceptability ratings of the intervention. In the pilot trial, participants will make these ratings after each session, in the open trial the ratings will be made pre and post intervention.
Arm/Group | Pilot Trial | Open Trial
All-Cause Mortality (participants affected / at risk) | 0/21 | 1/53
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/53
Other Adverse Events (participants affected / at risk) | 0/21 | 0/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot Trial (N=21) | Open Trial (N=53)
Serious, anticipated, unrelated adverse event (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/53/NCT03403153/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT03403153/ICF_001.pdf